CLINICAL TRIAL: NCT04439240
Title: MATCH Treatment Subprotocol W: Phase II Study of AZD4547 in Patients With Tumors With Aberrations in the FGFR Pathway
Brief Title: Testing AZD4547 as a Potential Targeted Treatment in Cancers With FGFR Genetic Changes (MATCH-Subprotocol W)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03213; NCI-2020-03213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-W (Other: ECOG-ACRIN Cancer Research Group); EAY131-W (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Plasma Cell Myeloma
Keywords: FGFR; AZD4547; NCI-MATCH
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — AZD4547

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (AZD4547) (Experimental): Patients receive AZD4547 PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: FGFR Inhibitor AZD4547

INTERVENTIONS:
Drug: FGFR Inhibitor AZD4547 — Given PO
  Other Names: AZD4547

SUMMARY:
This phase II MATCH treatment trial identifies the effects of AZD4547 in patients whose cancer has genetic changes called FGFR gene alterations. AZD4547 may stop the growth of cancer cells by blocking FGFR proteins which may be needed for cell growth. Researchers hope to learn if AZD4547 will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive FGFR inhibitor AZD4547 (AZD4547) orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have FGFR 1-3 mutation or translocation as determined by the MATCH screening assessment
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must have an echocardiogram (ECHO) or a nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have a left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients must have a pre-study eye exam by an ophthalmologist. Patients with current evidence of corneal or retinal disorder/keratopathy are excluded

Exclusion Criteria:

* Patients must not have known hypersensitivity to AZD4547 or compounds of similar chemical or biologic composition
* Patients must not have received prior FGFR specific inhibitors (e.g. BGJ398, erdafitinib, BAY1163877, LY2874455). Prior non-selective FGFR inhibitor treatment (e.g. pazopanib, dovitinib, ponatinib, brivanib, lucitanib, lenvatinib) will be allowed
* Patients must not have any history of or current evidence of renal or endocrine alterations of calcium/phosphate homeostasis, or history of or current evidence of extensive tissue calcification (by evaluation of the clinician), including but not limited to, the soft tissue, kidneys, intestine, myocardium and lung with the exception of calcified lymph nodes and asymptomatic vascular calcification per investigators' judgment
* Patients must not be currently using medications that can elevate serum phosphorous and/or calcium levels

  * Medications that increase serum calcium should be avoided. Over the counter calcium supplements, antacids that contain calcium (Tums) and vitamin D supplements (cholecalciferol and ergocalciferol) should be avoided. Prescription medications including lithium, hydrochlorothiazide and chlorthalidone must be used with caution
  * Medications that increase serum phosphate should be avoided. Over the counter laxatives that contain phosphate such as Fleets Oral or Fleets enema and Miralax should be avoided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young Kwang Chae, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Chae YK, Hong F, Vaklavas C, Cheng HH, Hammerman P, Mitchell EP, Zwiebel JA, Ivy SP, Gray RJ, Li S, McShane LM, Rubinstein LV, Patton D, Williams PM, Hamilton SR, Mansfield A, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of AZD4547 in Patients With Tumors Harboring Aberrations in the FGFR Pathway: Results From the NCI-MATCH Trial (EAY131) Subprotocol W. J Clin Oncol. 2020 Jul 20;38(21):2407-2417. doi: 10.1200/JCO.19.02630. Epub 2020 May 28. PMID 32463741
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7367548/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol W was activated on May 31, 2016. 70 patients were assigned to Subprotocol W after screening, all from screening cohort. Of the 70 patients, 52 patients from 47 different sites enrolled in the study between July 2016 and June 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For subprotocol W, patients had to have tumors harboring aberrations in FGFR 1-3.
Period: Overall Study
Arm/Group | Treatment (AZD4547)
Started | 52
Started Protocol Therapy | 50
Eligible | 49
Eligible and Started Protocol Therapy (2 patients ineligible, 1 patient never started treatment, 1 patient both ineligible and never started treatment. This is the primary analysis population.) | 48
Reported Adverse Events Data (1 of the 50 treated patients had no adverse events reported) | 49
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 52
Not completed — Ineligible | 2
Not completed — Never started treatment | 2
Not completed — Adverse Event | 12
Not completed — Death | 2
Not completed — Disease progression | 25
Not completed — Other diseases | 2
Not completed — Withdrawal by Subject | 3
Not completed — Clinical concerns for progression and increasing tumor marker | 1
Not completed — Symptomatic decline | 1
Not completed — Pogression of the lymphadenopathy | 1
Not completed — Clinical progression | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (AZD4547)
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 61 [22 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (AZD4547)
Number analyzed (Participants) | 48
percentage of participants | 8 [3 to 18]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. The 6-month PFS rate was estimated using the Kaplan-Meier method which can provide a point estimate for any specific time point. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS is determined
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (AZD4547)
Number analyzed (Participants) | 48
percentage of participants | 15 [8 to 31]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (AZD4547)
Number analyzed (Participants) | 48
months | 3.4 [1.8 to 4.7]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years
Description: All 52 patients enrolled to the trial were monitored for mortality. Of the 50 patients who received protocol therapy, 49 were evaluable for AEs (1 patient had no toxicity data)
Arm/Group | Treatment (AZD4547)
All-Cause Mortality (participants affected / at risk) | 44/52
Serious Adverse Events (participants affected / at risk) | 19/49
Other Adverse Events (participants affected / at risk) | 41/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (AZD4547) (N=49)
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 7
Small intestinal obstruction (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
GGT increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (AZD4547) (N=49)
Anemia (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 19
Alopecia (Skin and subcutaneous tissue disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 9
Nail discoloration (Skin and subcutaneous tissue disorders) | 7
Nail loss (Skin and subcutaneous tissue disorders) | 6
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 21
Dyspepsia (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 13
Hypercalcemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Dysgeusia (Nervous system disorders) | 10
Peripheral sensory neuropathy (Nervous system disorders) | 3
Blurred vision (Eye disorders) | 6
Dry eye (Eye disorders) | 12
Eye disorders - Other, specify (Eye disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT04439240/Prot_001.pdf